CLINICAL TRIAL: NCT01721200
Title: "Learning About Biologics"
Brief Title: "Learning About Biologics"-Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012-0294; 12-003011 (Other: Yale University)
Record Dates: First submitted 2012-10-10; First posted 2012-11-05 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; web based interactive learning tool
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Support Tool (Other): This study will examine the efficacy of a web-based educational decision support tool.
  Interventions: Other: Decision Support Tool
- Usual Care (Other): Usual Care Group will receive their biologic drug teaching from their rheumatologist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Decision Support Tool — Educational decision support tool for patients with rheumatoid arthritis
  Arms: Decision Support Tool
Other: Usual Care — Subjects randomized to the Usual Care Group will receive their biologic drug teaching from the rheumatologist as part of their routine care.
  Arms: Usual Care

SUMMARY:
This study is a randomized controlled trial designed to examine the efficacy of an educational decision support tool for patients with rheumatoid arthritis who continue to have active disease despite use of traditional disease modifying drugs. The study will take place at Geisinger Medical Center in Danville, PA. Eligible subjects will be identified by the treating physician and those providing consent will be randomized to usual care versus use of the decision support tool.

DETAILED DESCRIPTION:
Data suggest that undertreatment of rheumatoid arthritis (RA) patients may be in part due to inadequate decision support when they face whether or not to start biologic therapy. No proven way exists to inform or support RA patients who are candidates for biologic therapy. Communicating information about biologic medication is particularly challenging because of the sheer number of risks to disclose, the difficulty explaining the risks of extremely rare adverse events (AEs), and the tendency for people to discount (or underweight) future benefits.

Dr Liana Fraenkel at Yale University is the Primary Investigator and developer of this theory-based high quality decision support tool to effectively inform RA patients who are candidates for biologics. Dr. Eric Newman will be Principal Investigator for the project which will be conducted at Geisinger Medical Center. All subjects enrolled will complete a baseline survey and then will be randomized to use of the decision support tool or to usual care. Those randomized to usual care will be offered the opportunity to access the tool once enrollment is closed and all follow-up visits have been completed.

Outcomes will be assessed at two and six weeks after the baseline visit by the Geisinger Telephone Survey and Interviewing Facility. This facility is equipped with 12 computers and runs two shifts a day. The Survey Unit uses a state-of-the-art Windows based Computer Assisted Telephone Interview (CATI) system to administer surveys and collect research data. The group holds 12 interviewer licenses for the CATI system. Trained and experienced interviewers are available to make the calls from 9 am to 9 pm Monday through Friday and from 10 am to 2 pm on Saturdays.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Able to speak and read English
* Meet the revised American College of Rheumatology criteria for the diagnosis of RA
* Have active disease warranting initiation of a new biologic (or small molecule if and when FDA-approved) therapy as determined by their rheumatologist

Exclusion Criteria:

* Fail to meet the inclusion criteria
* Have a current infection
* Have cancer of any type diagnosed within the past five years (except non-melanoma skin cancer)
* Have a history of lymphoma, leukemia, or melanoma
* Have a chronic inflammatory disease (in addition to rheumatoid arthritis) requiring treatment with immunosuppressive medications
* Have chronic liver disease due to hepatitis C or B
* Are HIV positive
* Have a positive screening test for tuberculosis (tuberculin skin test or interferon-gamma release assay) or radiographic lesions suggestive of inactive tuberculosis and have not completed an adequate course of chemoprophylactic therapy
* Are hearing or visually impaired
* Are scheduled for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liana Fraenkel, MD, MPH, Principal Investigator — Yale University
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fraenkel L, Matzko CK, Webb DE, Oppermann B, Charpentier P, Peters E, Reyna V, Newman ED. Use of Decision Support for Improved Knowledge, Values Clarification, and Informed Choice in Patients With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2015 Nov;67(11):1496-502. doi: 10.1002/acr.22659. PMID 26195173
- See also: Geisinger Health System — http://www.geisinger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were RA patients currently being treated by one of six rheumatologists practicing in the Geisinger Rheumatology Department in Danville, Pennsylvania who were at least 18 years of age, able to speak and read English & had active disease warranting initiation, or change, of a biologic therapy as determined by their treating rheumatologist.
Pre-assignment Details: Subjects excluded if hearing or visually impaired; scheduled for surgery;current infection; cancer past five years (except non-melanoma),lymphoma, leukemia,melanoma;chronic inflammatory disease (+ RA) immunosuppressive RX; chronic liver disease, hepatitis C or B;HIV +; TB+x-ray lesions of inactive TB & no chemoprophylactic therapy..
Period: Overall Study
Arm/Group | Decision Support Tool | Usual Care
Started | 62 | 63
Completed 2 Week Follow-up | 60 | 61
Completed | 59 | 58
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Population: 152 subjects approached. out of this number 125 patients agreed to participate and were randomized.
  125 subjects completed baseline survey. 63 were randomized to control group and 62 to intervention. 61 completed two week follow-up survey in control group and 60 in intervention group.
  58 completed 8 week survey and 59 in intervention group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Support Tool | Usual Care | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 63 | 125
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.3) | 56.2 (11.4) | 55.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 44 | 85
  Male | 21 | 19 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 59 | 59 | 118
  More than one of the above races | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Are Classified as Having Made an Informed Value Concordant Choice at 2 Weeks
Description: We classified subjects as having made an informed choice to escalate care if they answered at least 75% of the knowledge questions correctly and had low decisional conflict as defined by a score of 25 or lower on the combined subjective knowledge and values clarity subscales.
Time Frame: 2 weeks
Measure: Number; unit: Percentage of subjects
Groups:
- Intervention Group: Randomized to view the decision support tool.
- Control: Usual Care
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 60 | 61
Percentage of subjects | 32 | 13

2. Secondary Outcome: Patient-physician Communication
Description: Patient-physician communication will be measured using the COMRADE (Combined Outcome Measure for Risk communication And treatment Decision making Effectiveness): a 20-item scale composed of two subscales which address the quality of risk communication (process measure) and the quality of the decision making process (outcome measure). Items are measured on a 5-point agree scales. The COMRADE is a includes two sub-scales (each composed of 10 items): one for risk communication (a process measure) and a second for confidence in decision (an outcome measure). Subscales are summed to generate a total score (Range 20-100). Higher scores reflect poorer outcomes.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Intervention | Control
Number analyzed (Participants) | 59 | 58
units on a scale | 35.8 (12.2) | 35.6 (11.3)

3. Secondary Outcome: Use of Biologics
Description: Use of biologics: The number of patients received a prescription for a new biologic by eight weeks.
Time Frame: 8 weeks
Measure: Number; unit: Number of subjects
Arm/Group | 1 Intervention | Control
Number analyzed (Participants) | 60 | 61
Number of subjects | 51 | 49

4. Secondary Outcome: To Test Screening and Recruitment Procedures
Description: To test screening and recruitment procedures we will measure the number of eligible patients, the number of patients excluded by each exclusion criterion, the number of patients referred by rheumatologists each week, and the proportion of patients who agree to participate.
Time Frame: 8 weeks
Population: Data not collected
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Test Uptake
Description: To test uptake and adherence to the intervention we will measure the proportion of patients randomized to the intervention who access the tool, complete the Best Worse Scaling exercise, print a handout, and use the handout during a follow-up visit with their rheumatologist (for subjects having a second visit within eight weeks). Note, subjects without access to a printer will have the opportunity to do so in the office.
Time Frame: 8 weeks
Population: Data not collected
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Acceptability to Physicians
Description: Acceptability to physicians will be assessed using four items coded on 5-point Frequency scales (1= None of the time and 5= All of the time) administered by the research assistant once all patient follow-up interviews have been completed:
  1. Did the tool make it easier to talk about treatment with your patients?
  2. Did the tool increase the amount of time you spent discussing therapy with your patients?
  3. Did the tool decrease the amount of time you spent discussing therapy with your patients?
  4. Did the tool improve the quality of informed consent for patients initiating biologics?
Time Frame: 8 weeks
Population: Data not collected
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

7. Secondary Outcome: To Test Adherence to the Intervention
Description: The session management system will record the time spent on each module visited within the tool to assess adherence.
Time Frame: 8 weeks
Population: These data were not collected.
Arm/Group | Usual Care | Decision Support Tool
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Changes in Knowledge
Description: Knowledge will be measured using the 20 True/False statements developed for the initial pre-post test study. The number of correct responses are summed to yield a knowledge score (possible range= 0-20). The item order was determined using a random-numbers generator.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 1 Intervention | Control
Number analyzed (Participants) | 62 | 63
units on a scale | 1 [-1 to 2] | 0 [-2 to 1]

9. Secondary Outcome: Changes in Willingness
Description: Willingness: Patients' propensity towards biologics will be measured using the choice predisposition scale (65): This item is coded on a 11-point scale anchored by "Not willing at all" and "Extremely willing" with "Unsure" at the midpoint (65). Higher scores reflect greater willingness.
Time Frame: 8 weeks
Population: Follow-up data not collected because of ceiling effect.
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Changes in Perceived Knowledge
Description: Perceived knowledge and value clarity will be measured using two subscales from the well-validated Decisional Conflict Scale (66). Each subscale is composed of 3 items measured on 5-point agree scales. Scores are rescaled to range from 0 to 100. Higher scores reflect greater conflict (poorer outcomes).
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 59 | 58
units on a scale | -16.7 [-33 to 0] | -8.3 [-25 to 8.3]

ADVERSE EVENTS:
Arm/Group | Usual Care | Decision Support Tool
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No